CLINICAL TRIAL: NCT01741831
Title: Regulatory Post Marketing Surveillance of Prezista 400mg Tablet
Brief Title: A Post Marketing Survey Study to Evaluate the Safety and Effectiveness of Prezista
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100805; TMC114HIV4074 (Other: Janssen Korea, Ltd., Korea); Prezista PMS (Other: Janssen Korea, Ltd., Korea); DRV-C-11-KR-001-V06 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Acquired Immune Deficiency Syndrome
Keywords: Acquired Immune Deficiency Syndrome; AIDS; TMC114; Darunavir; Prezista
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Darunavir: Patients having Acquired Immune Deficiency Syndrome (AIDS) will be taking darunavir as per recommended doses.
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Darunavir will be administered as per the recommended doses and will be given orally for a period of 24 weeks. For treatment naive (never received treatment for AIDS) patients: Darunavir 800 mg will be adminstered along with ritonavir 100 mg once daily. For experienced patients: Darunavir 600 mg will be administered along with ritonavir 100 mg twice daily.
  Other Names: Prezista

SUMMARY:
The purpose of this study is to assess the safety data of darunavir in a natural clinical practice.

DETAILED DESCRIPTION:
This is a non-interventional (a scientific study to make a clear and easy understanding of the cause and effect relationship), prospective (in which the participants are first identified and then followed forward as time passes), consecutive survey for collecting safety and efficacy data of darunavir in treatment of Acquired Immune Deficiency Syndrome (AIDS) in a natural clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are prescribed with darunavir for treatment of Acquired Immune Deficiency Syndrome (AIDS)

Exclusion Criteria:

* Known hypersensitivity to Prezista
* Prezista coadministered with medicinal products that are highly dependent on CYP3A for clearance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients who are diagnosed with Acquired Immune Deficiency Syndrome (AIDS), and who are prescribed with darunavir for treatment of AIDS.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2012-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | Up to 30 days from end of treatment

SECONDARY OUTCOMES:
Number of patients with viral load | Screening, Week 12, Week 24
Number of patients with CD4 T-cell count | Screening, Week 12, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (1):
- Daegu, South Korea